CLINICAL TRIAL: NCT06963190
Title: Impact of Inspiratory Muscle Training (IMT) With Intermittent Variable Resistance (IVR) Versus Constant Resistance (CR) on Functional Capacity in Lung Transplantation (LTx) Patients
Brief Title: Impact of Inspiratory Muscle Training (IMT) With Intermittent Variable Resistance (IVR) Versus Constant Resistance (CR) on Functional Capacity in Lung Transplantation (LTx) Patients (I-TRAIN-LTx Study)
Acronym: I-TRAIN-LTx
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Marqués de Valdecilla (Other)
Responsible Party: Principal Investigator, Andrea Pérez Zabaleta, Principal investigator, Hospital Universitario Marqués de Valdecilla
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Impact of IMT en LTX patients
Record Dates: First submitted 2025-03-16; First posted 2025-05-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Lung Transplantation
Keywords: Respiratory Muscle Training; Lung Transplantation; Respiratory Function Tests; Spirometry; Blood Gas Analysis; Walk Test; Diaphragm Paralysis
MeSH Terms: conditions — Respiratory Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Constant Resistance (CR) (Active Comparator)
  Interventions: Other: Constant Resistance (CR)
- Intermittent Variable Resistance (IVR) (Experimental)
  Interventions: Other: Intermittent Variable Resistance (IVR)

INTERVENTIONS:
Other: Constant Resistance (CR) — Will perform inspiratory muscle training at 30% of MIP. Two daily sessions of 30 breaths or 10 minutes.
  Arms: Constant Resistance (CR)
Other: Intermittent Variable Resistance (IVR) — Will perform inspiratory muscle training at 30% of MIP. This will consist of two daily sessions of 30 breaths or 10 minutes. Additionally, the participant will complete 8 sets of 3 repetitions at 60% of the MIP, distributed throughout the day, with a one-minute rest between each repetition.
  Arms: Intermittent Variable Resistance (IVR)

SUMMARY:
- Objectives: Primary Objective: To compare Maximum Inspiratory Pressure (MIP) in lung transplant (LT) patients between the use of inspiratory muscle training (IMT) with intermittent variable resistance (IVR) or constant resistance (CR) during the first six months post-transplant.

Secondary Objectives: To determine whether there are differences in the outcomes of IMT with IVR and IMT with CR in the six-minute walk test, spirometry values, and arterial blood gas analysis within the first six months post-transplant.

To analyze the influence of relevant clinical conditions on dependent variables in both groups: duration of mechanical ventilation during the immediate postoperative period of LT and presence of diaphragmatic paralysis.

To analyze the proportion of patients with Baseline Lung Allograft Dysfunction (BLAD) in both intervention groups.

- Methodology: Design: Open-label, two-arm, randomized clinical trial.

Intervention: Random allocation into:

CR Group: Will perform IMT at 30% of MIP. IVR Group: Will perform IMT at 30% and 60% of MIP.

Population and Sample: Patients undergoing lung transplantation.

Demographic and LT-related variables: Sex, date of birth, height, weight, body mass index, type of transplant, underlying disease leading to transplantation, phrenic paralysis, length of stay in the intensive care unit, days on mechanical ventilation, primary graft dysfunction, and acute rejection.

Dependent Variables: MIP, spirometry, arterial blood gas analysis, six-minute walk test, and BLAD criteria.

DETAILED DESCRIPTION:
Background and Current State of Knowledge

According to the World Health Organization, chronic obstructive pulmonary disease (COPD) is the fourth leading cause of death worldwide, accounting for 3.5 million deaths in 2021, approximately 5% of all global fatalities.

Lung transplantation (LT) is a treatment option for patients with severe, irreversible, non-neoplastic chronic respiratory diseases when all other therapeutic options have been exhausted, provided that post-transplant survival and quality of life are superior to those of the underlying condition.

The International Society for Heart and Lung Transplantation (ISHLT) has recorded over 70,000 lung transplants worldwide since its registry began. In recent years, the number of annual lung transplants has increased significantly.

In Spain, a global leader in organ donation and solid organ transplantation in 2023, 479 lung transplants were performed, according to the Spanish National Transplant Organization (ONT). The main indications for lung transplantation were COPD (40%), diffuse interstitial lung disease (DILD) (36%), and other conditions (24%), including retransplantation, cystic fibrosis, bronchiectasis, and pulmonary hypertension.

Patients with COPD and DILD, the most common indications for lung transplantation, experience exercise intolerance, dyspnea, and decreased respiratory muscle strength and endurance-symptoms that worsen post-transplant. Newly transplanted patients have denervated lungs, a lack of cough reflex, and reduced mucociliary clearance due to factors such as mechanical ventilation, anesthesia, or immunosuppressive medications. These factors may contribute to early complications, including atelectasis and secondary infections, which require treatment through respiratory physiotherapy.

The diaphragm is the primary inspiratory muscle, and diaphragmatic dysfunction can involve partial or total loss of function, affecting one or both hemidiaphragms. Main issues include reduced muscle strength, endurance alterations, limited mobility, and diaphragmatic fatigue.

In COPD patients, diaphragmatic structural changes include negative alterations and adaptive modifications, directly impacting diaphragm function and its ability to meet respiratory demands.

Among the negative changes, diaphragmatic atrophy is prominent, with a 30% reduction in myosin heavy chain content in mild-to-moderate COPD patients and a 30%-40% decrease in muscle fiber cross-sectional area in severe cases. This leads to loss of contractile strength, elasticity, and functionality.

Conversely, adaptive changes occur in response to increased respiratory demand, notably the transformation of type II muscle fibers into type I fibers, which are more fatigue-resistant and have a predominantly oxidative metabolism. However, despite enhancing endurance, these adaptations reduce total diaphragmatic strength, as type I fibers generate less force than type II fibers.

Idiopathic pulmonary fibrosis (IPF), the most common form of DILD, shares similarities with COPD in terms of exercise limitation due to dyspnea. Studies show reduced diaphragmatic mobility during deep breathing and greater muscle weakness in IPF patients compared to healthy individuals.

Although chronic lung allograft dysfunction (CLAD) remains the primary cause of post-transplant mortality, a newly described phenomenon called Baseline Lung Allograft Dysfunction (BLAD) is characterized by an inability to achieve FEV1 and/or FVC values above 80%. Although its causes remain unclear, alterations in MIP may be related.

Several studies on IMT in COPD and IPF patients, as well as post-cardiac surgery patients, conclude that IMT is beneficial in reducing dyspnea, improving muscle strength and endurance, increasing exercise capacity, and enhancing quality of life.

MIP is determined by performing a maximal inspiration from residual volume under static conditions, assessing diaphragm strength. However, no consensus exists on the required load to strengthen the diaphragm. Training loads vary from 30% to 60% of MIP, with most protocols recommending 10-15 minutes twice daily at a constant load.

Few studies have examined IMT in recently transplanted patients. A 2024 review by Polastri et al. analyzed 64 lung transplant candidates and recipients, showing that participants used a threshold valve device with resistance levels between 30% and over 50% of MIP, training twice daily with 30-60 inspirations or for 15 minutes. A 2022 pilot study by Graur et al. found significant improvements in MIP and six-minute walk test results in transplanted patients performing IMT. Training intensity progressively increased from 15% to 60% of MIP within the first month. Most other studies have small sample sizes or focus on lung transplant candidates or heart-lung transplant recipients.

Hypothesis

Primary Hypothesis: IMT with IVR has a greater impact on functional capacity than IMT with CR in lung transplant patients in the short and medium term.

Secondary Hypotheses:

IMT with IVR significantly improves MIP, six-minute walk test results, spirometry values, and arterial blood gas levels compared to IMT with CR in lung transplant patients in the short and medium term.

Patients requiring longer mechanical ventilation durations and those with diaphragmatic paralysis will benefit more from IMT with IVR than IMT with CR.

The proportion of BLAD patients will be lower in the IVR group than in the CR group.

Ethical Considerations The study will be approved by the Ethics Committee for Drug Research (CEIm). Patients will provide written informed consent, adhering to EU Regulation 2016/679 (GDPR) and Spanish Organic Law 3/2018 on data protection. The study follows the Declaration of Helsinki and Good Clinical Practices (GCP) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years) who has undergone lung transplantation (single-lung or double-lung) at our center.
* Alert and cooperative (Glasgow Coma Scale >13 points).
* Hemodynamically stable (blood pressure between 90/60 and 165/90 mmHg; heart rate between 60 and 130 beats per minute).
* No disabling dyspnea at rest (maintained at mild levels according to the Borg scale or NYHA class I-II), even if requiring supplemental oxygen with a saturation >89%.
* No limiting chest pain interfering with respiratory therapy.

Exclusion Criteria:

* Patients unable to cooperate with treatment due to lack of necessary instrumental cognitive skills.
* Perceived non-adherence to pharmacological and non-pharmacological treatment by healthcare personnel.
* Need for continuous non-invasive mechanical ventilation, high-flow oxygen therapy, or Venturi mask.
* Patients with significant neurological disorders, severe polyneuropathies, or stroke (CVA).
* Presence of tracheostomy, active hemoptysis, bronchial suture dehiscence.
* Significant air leak with clinical repercussions.
* Any clinical condition that, in the investigator's judgment, poses a risk to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-31 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dependent variables | Measurements will be performed at the time of recruitment (baseline) and at months 1, 2, 4, and 6 post-transplant.
  Maximal inspiratory pressure: Expressed in cmH₂O.
Dependent variables | Measurements will be performed at the time of recruitment (baseline) and at months 1, 2, 4, and 6 post-transplant.
  Spirometry: Forced expiratory volume in the first second (FEV1) in mL and percentage of predicted, forced vital capacity (FVC) in mL and percentage, and FEV1/FVC ratio.

SECONDARY OUTCOMES:
Demographic and Transplant-Related Variables | Measurements will be performed at the time of recruitment (baseline)
  Length of stay in the intensive care unit (ICU) (days)
Demographic and Transplant-Related Variables | Measurements will be performed at the time of recruitment (baseline)
  Duration of mechanical ventilation (days)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Marqués de Valdecilla, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No